CLINICAL TRIAL: NCT04379739
Title: Neoadjuvant Camrelizumab Plus Apatinib or Platinum-based Chemotherapy for Potentially Resectable (Resectable and Initially Unresectable) II-III Non-small Cell Lung Cancer
Brief Title: Neoadjuvant PD-1 Antibody Plus Apatinib or Chemotherapy for Non-small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Peng Zhang, Director of thoracic department, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-NSCLC-II-001 (LungMate-003)
Record Dates: First submitted 2020-04-19; First posted 2020-05-07 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — camrelizumab; apatinib; Platinum Compounds

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- camrelizumab + apatinib (Experimental): Neoadjuvant treatment stage: camrelizumab 200mg, q3w, i.v., 2-4 cycles; apatinib 250 mg, qd, p.o. 3 weeks per cycle, 2-4 cycles, then receive chest CT evaluation.
  Surgery stage: the patients will receive radical surgery 3-4 weeks after the neoadjuvant treatment.
  Adjuvant treatment stage: according to the NCCN guidelines.
  Interventions: Drug: Camrelizumab
- camrelizumab + platinum-based chemotherapy (Experimental): Neoadjuvant treatment stage: camrelizumab 200mg, q3w, i.v., 2-4 cycles; platinum-based chemotherapy (squamous: carboplatin AUC5, gemcitabine 1000mg/m2; non-squamous: carboplatin AUC5, pemetrexed 500mg/m2) q3w, i.v., 2-4 cycles, then receive chest CT evaluation.
  Surgery stage: the patients will receive radical surgery 3-4 weeks after the neoadjuvant treatment.
  Adjuvant treatment stage: according to the NCCN guidelines.
  Interventions: Drug: Camrelizumab

INTERVENTIONS:
Drug: Camrelizumab — camrelizumab 200mg, q3w, i.v., 2-4 cycles;
  Other Names: Apatinib; Platinum-based chemotherapy

SUMMARY:
Immunotherapy with anti-programmed death 1 (PD-1) antibodies has revolutionized the treatment of metastatic and advanced NSCLC, but its application in neoadjuvant setting has not been well established. Results from a pilot clinical study reported the safety and feasibility of neoadjuvant PD-1 blockade. There are several neoadjuvant immunotherapy (NEOSTAR, LCMC3, NADIM, IMpower131) ongoing, and the preliminary results are reported in 2019 American Society of Clinical Oncology, which show promising therapeutic prospect. However, the therapeutic response rate (major pathologic response [MPR]) are not so good (20% - 45%) for PD-1 inhibitor monotherapy. To improve the therapeutic response, the investigators design a multiple-canter, open-label, phase II trial for stage II-III potentially resectable (resectable and initially unresectale) NSCLC. The participants will receive neoadjuvant PD-1 inhibitor (camrelizumab) combined with antiangiogenic drug (apatinib) or platinum-based chemotherapy.

DETAILED DESCRIPTION:
Detailed Description:

This is a multiple-canter, open-label, phase II trial, 2-4 cycles treatment will be planned as neo-adjuvant therapy for NSCLC participants in stage II-III.

Study design:

Participants: Newly diagnosed Resectable and Initially Unresectale II-III NSCLC without EGFR/ALK mutation.

Treatment:

Group A：camrelizumab 200 mg q3w i.v. for 2-4 cycles, platinum-based chemotherapy q3w i.v for 2-4 cycles before surgery.

Group B：camrelizumab 200 mg q3w i.v. for 2-4 cycles, apatinib 250mg qd po 3w/cycle for 2-4 cycles before surgery;

Endpoints:

Primary objectives are to assess MPR and safety. Secondary objective is to assess 2-year overall survival (OS), disease-free survival (DFS), OS etc.

Exploratory end point is to explore biomarkers.

ELIGIBILITY:
Inclusion Criteria:

Group A:

1. Aged 18-75 years;
2. Eastern Cooperative Oncology Group (ECOG) performance-status score of 0 or 1;
3. Histological or cytological diagnosis of NSCLC by needle biopsy, and clinical stage II-III according to the TNM classification (8th edition) validated by radiological examination or EBUS;
4. At least 1 measurable lesion according to RECIST 1.1;
5. Life expectancy is at least 12 weeks;
6. Adequate hematological function, liver function and renal function:

   * Hemoglobin ≤ 90 g/L (which can be maintained or exceeded by blood transfusion);
   * Absolute neutrophil count (ANC) ≤ 1.5 *10^9/L;
   * Platelet count ≤ 100 * 10^9/L;
   * Total bilirubin ≤ 1.5 times of upper limit of normal (ULN);
   * Alanine glutamate transaminase (ALT), straw glutamate transaminase (AST) and alkaline phosphatase (ALP) ≤ 2.5 * ULN;
   * Creatinine ≤ 1.5 * ULN, Creatinine clearance rate ≤ 60ml/min;
   * The international standardized ratio of prothrombin time (INR) ≤ 1.5 R in patients who have not received anticoagulation therapy, and the partial thrombin time (APTT) ≤ 1.5 * ULN.
7. Without systemic metastasis (including M1a, M1b and M1c);
8. With the expectation of radical surgery therapy, or with the expectation of complete resection after treatment;
9. Patients with normal lung function can tolerate surgery;
10. The child-bearing female must undergo pregnancy test (serum or urine) within 72 hours before drug administrating and the result shall be negative. Reliable contraceptive measures, such as intrauterine device, contraceptive pill and condom, shall be adopted during the trial and within 90 days after the last dosage of the drug. The male participants whose partners are child-bearing shall use condom for contraception during the trial and within 30 days after completion of the trial;
11. Signed and dated informed consent.

Group B:

1. Aged 18-75 years;
2. Eastern Cooperative Oncology Group (ECOG) performance-status score of 0 or 1;
3. Histological or cytological diagnosis of NSCLC by needle biopsy, and clinical stage II-III according to the TNM classification (8th edition) validated by radiological examination or EBUS;
4. Enough tumor samples from biopsy to testing PD-L1 expression level, and PD-L1 ≥ 1%
5. At least 1 measurable lesion according to RECIST 1.1;
6. Life expectancy is at least 12 weeks;
7. Adequate hematological function, liver function and renal function:

   * Hemoglobin ≤ 90 g/L (which can be maintained or exceeded by blood transfusion);
   * Absolute neutrophil count (ANC) ≤ 1.5 *10^9/L;
   * Platelet count ≤ 100 * 10^9/L;
   * Total bilirubin ≤ 1.5 times of upper limit of normal (ULN);
   * Alanine glutamate transaminase (ALT), straw glutamate transaminase (AST) and alkaline phosphatase (ALP) ≤ 2.5 * ULN;
   * Creatinine ≤ 1.5 * ULN, Creatinine clearance rate ≤ 60ml/min;
   * The international standardized ratio of prothrombin time (INR) ≤ 1.5 R in patients who have not received anticoagulation therapy, and the partial thrombin time (APTT) ≤ 1.5 * ULN.
8. Without systemic metastasis (including M1a, M1b and M1c);
9. With the expectation of radical surgery therapy, or with the expectation of complete resection after treatment;
10. Patients with normal lung function can tolerate surgery;
11. The child-bearing female must undergo pregnancy test (serum or urine) within 72 hours before drug administrating and the result shall be negative. Reliable contraceptive measures, such as intrauterine device, contraceptive pill and condom, shall be adopted during the trial and within 90 days after the last dosage of the drug. The male participants whose partners are child-bearing shall use condom for contraception during the trial and within 30 days after completion of the trial;
12. Signed and dated informed consent.

Exclusion Criteria:

Group A:

1. The patient has undergone any systemic anti-cancer treatment for NSCLC, including surgical treatment, local radiotherapy, cytotoxic drug treatment, targeted drug treatment, immunotherapy or Chinese medicine treatment, etc. (excluding the malignant tumors that were resected radically and did not recurrent more than 5 years);
2. Non-squamous cell carcinoma with EGFR active mutation positive or ALK rearrangement;
3. The patient suffered from other cancers (except cervical carcinoma in situ, cured basal cell carcinoma and bladder epithelial tumor [including Ta and Tis]) within 5 years before the enrollment;
4. The patient suffers from any active autoimmune disease or have the history of autoimmune disease, such as uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism (can be included after hormone replacement therapy), tuberculosis; Note: The patients with complete remission of childhood asthma and without any interventions in adult life could be included. The patients with skin diseases (like vitiligo, psoriasis or alopecia) who do not need systematic therapy could be included.
5. Suffering or having the history of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiological pneumonia, drug-induced pneumonia, radiologically confirmed active pneumonia, or severe impairment of lung function;
6. Participants who were systemically treated with corticosteroids (prednisone or other corticosteroids >10 mg/ day) or other immunosuppressive agents within 2 weeks prior to first administration. In the absence of active autoimmune disease, inhaled or topical corticosteroids and adrenal hormone replacement therapy with a dose of less than 10 mg/ day of prednisone are permitted;
7. Allergy to the test drug;
8. The patient is a carrier of active hepatitis B, hepatitis C or HIV;
9. Pregnancy or breast-feeding women; child-bearing participants who could not or are unwilling to take contraceptive measures.
10. Patients with eurological or psychiatric disorders history were lack of treatment compliance;
11. Other situations in which investigators thought the patients not suit to be included.

Group B:

1. The patient has undergone any systemic anti-cancer treatment for NSCLC, including surgical treatment, local radiotherapy, cytotoxic drug treatment, targeted drug treatment, immunotherapy or Chinese medicine treatment, etc. (excluding the malignant tumors that were resected radically and did not recurrent more than 5 years);
2. Non-squamous cell carcinoma with EGFR active mutation positive or ALK rearrangement;
3. The patient suffered from other cancers (except cervical carcinoma in situ, cured basal cell carcinoma and bladder epithelial tumor [including Ta and Tis]) within 5 years before the enrollment;
4. The patient suffers from any active autoimmune disease or have the history of autoimmune disease, such as uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism (can be included after hormone replacement therapy), tuberculosis; Note: The patients with complete remission of childhood asthma and without any interventions in adult life could be included. The patients with skin diseases (like vitiligo, psoriasis or alopecia) who do not need systematic therapy could be included.
5. Suffering or having the history of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiological pneumonia, drug-induced pneumonia, radiologically confirmed active pneumonia, or severe impairment of lung function;
6. Participants who were systemically treated with corticosteroids (prednisone or other corticosteroids >10 mg/ day) or other immunosuppressive agents within 2 weeks prior to first administration. In the absence of active autoimmune disease, inhaled or topical corticosteroids and adrenal hormone replacement therapy with a dose of less than 10 mg/ day of prednisone are permitted;
7. Imaging (CT or MRI) shows that the tumor has invaded or blurred the boundary with the great vessels;
8. The participants who suffered thrombus events, such as stroke (including temporary ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism;
9. Having clinically significant bleeding symptoms or had definite bleeding tendency, such as gastrointestinal bleeding or bleeding ulcer, or were receiving thrombolytic therapy or anticoagulant therapy within 3 months before enrollment;
10. Having symptoms of obvious hemoptysis or daily hemoptysis of 2.5ml or more within 1 month before enrollment;
11. Participants with hypertension and unable to obtain good control with antihypertensive drugs (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg); Grade II or larger myocardial ischemia or myocardial infarction, poorly controlled arrhythmia (including QTc interphase, male ≥ 450ms, female ≥ 470ms); According to NYHA, grade Ⅲ ~ Ⅳ cardiac insufficiency, or left ventricular ejection fraction (LVEF) < 50%;
12. The participants have undergone other major systemic operations or suffered from severe trauma within 2 months before the enrollment;
13. Urinary protein ≥ ++, or urinary protein ≥1g at 24h or severe liver and kidney dysfunction;
14. Uncontrollable pleural effusion, pericardial effusion or ascites requiring repeated drainage;
15. Allergy to the test drug;
16. The patient is a carrier of active hepatitis B, hepatitis C or HIV;
17. Pregnancy or breast-feeding women; child-bearing participants who could not or are unwilling to take contraceptive measures.
18. Patients with eurological or psychiatric disorders history were lack of treatment compliance;
19. Other situations in which investigators thought the patients not suit to be included.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2020-07-26 (Actual); Primary Completion 2022-06-29 (Actual); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Major pathologic response (MPR) | up to 5 months
  MPR is defined as the proportion of participants who have achieved major pathologic response (on routine hematoxylin and eosin staining, tumors with no more than 10% viable tumor cells) in all participants who have completed the neoadjuvant therapy before surgery.

SECONDARY OUTCOMES:
2-year OS | up to 27 months
  It is defined as the time from enrollment to death of participant due to any cause in 2 years. In the case of a patient who still survives at the time of analysis, the date of last contact will be taken as the censoring date.
Objective response rate (ORR) | up to 4 months
  It refers to the proportion of patients who have had a complete response or partial response (according to RECIST1.1) as confirmed by CT evaluation after 3 weeks in all patients who have completed the neoadjuvant therapy. Only patients with measurable lesions at baseline will be analyzed.
Disease-free survival (DFS) | up to 60 months
  It refers to the time from radical surgery to relapse or death of a participant due to disease progression. In the case of a patient who still survives at the time of analysis, the latest evaluation date will be used for interpolation (censoring).
Overall survival (OS) | up to 63 months
  It is defined as the time from enrollment to death of participant due to any cause. In the case of a patient who still survives at the time of analysis, the date of last contact will be taken as the censoring date. In the event of a patient with the survival status unknown, the date when the patient is last known to be alive will be used for interpolation (censoring).
Safety: frequency of severe adverse events | up to 6 months
  The frequency of severe adverse events from the participants enrolling to 90 days after the last drug administration or 30 days after surgery or new anti-cancer therapy, which comes first.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shang'ai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
The researchers will consider whether IPD is available to other researchers only after the paper is published.

REFERENCES:
- [Derived] Ji S, Sheng Z, Bian D, Bao M, Jin K, Zhang W, Zhu X, Sun F, Xia H, Zhang H, Shen Z, Yu H, Zhang L, Huang J, Peng Z, Song N, Wang H, Qian B, Zhu Y. Neoadjuvant camrelizumab plus chemotherapy or apatinib for resectable stage IIA-IIIA NSCLC: a multicenter, two-arm, phase II exploratory trial. BMC Med. 2025 Jul 18;23(1):429. doi: 10.1186/s12916-025-04250-4. PMID 40682106